CLINICAL TRIAL: NCT00816374
Title: Tailored Intervention for Melanoma Patient's Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FCCC- 05-805; IRB 05-805
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma
Keywords: cutaneous malignant melanoma; CMM; total cutaneous examination; TCE; skin self-examination; SSE; first degree relatives; FDR; skin cancer protection; skin cancer screening
MeSH Terms: conditions — Melanoma; Melanoma, Cutaneous Malignant | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Group I
  Interventions: Other: Reading materials and discussions; Other: Questionnaires
- 2 (Other): Group II
  Interventions: Other: Reading materials and discussions; Other: Questionnaires

INTERVENTIONS:
Other: Reading materials and discussions — We will send 3 sets of materials via mail, containing information about melanoma prevention and detection, 1 set each month for 3 months. Materials published by:
  * The American Cancer Society
  * The American Academy of Dermatology
  * The Skin Cancer Foundation
  The pamphlets contain information about ways to reduce risk for skin cancer including:
  * Sun protection practices
  * Risk factors for melanoma
  * Information about what melanoma looks like
  * How to do skin self-examinations
  There will also be a telephone discussion with a health educator, discussing melanoma and other information contained in the pamphlets.
  Other Names: Supportive Care Intervention; Behavioral
  Arms: 1
Other: Reading materials and discussions — We will send 3 separate pamphlets created specifically for participants. We will send 1 pamphlet each month for 3 months. The information in the pamphlets will be based on answers from the first survey. These pamphlets will contain information about:
  * Melanoma and skin cancer protection guidelines
  * The benefits of skin screening practices
  * Ways to protect yourself from the sun
  In addition to these pamphlets, there will be a telephone discussion with a health educator to discuss melanoma and other information contained in the pamphlets.
  Other Names: Supportive Care Intervention; Behavioral
  Arms: 2
Other: Questionnaires — Both groups will complete 3 surveys; at the beginning, 3 months later, 6 months after the second survey. Each survey will ask about:
  * knowledge of melanoma
  * current and past skin cancer screening practices
  * current and past sun protection practices
  * attitudes about skin cancer and sun protection
  * feelings about relative's melanoma diagnosis and treatment
  Other Names: Supportive Care Intervention; Behavioral

SUMMARY:
The purpose of the investigators' study is to find the best way to provide information about sun protection and skin cancer detection. The investigators want to see which of two methods most improves sun protection and screening attitudes and practices. The investigators hope to improve these attitudes and practices among people who are at higher risk for melanoma. People at higher risk for melanoma are first degree relatives (mother, father, sibling or child) of people diagnosed with melanoma.

DETAILED DESCRIPTION:
Eligible patients will be contacted to find out whether they have any living first degree relatives that we may contact to discuss their participation in our study.

Eligible first degree relatives (FDRs) will participate in our study as outlined under Interventions.

ELIGIBILITY:
Inclusion Criteria - Patients (for referral of FDRs):

* Newly diagnosed with cutaneous malignant melanoma (CMM) within the past 2 years but more than 3 months prior to being approached
* Seen at FCCC, FCCC Network, Temple, MCC, or HUP patient clinics
* Greater than 18 years of age
* English speaking
* Able to give meaningful informed consent
* Does NOT have a first-degree relative with CMM

Inclusion Criteria - FDR (First Degree Relative):

* Current age of at least 21 years
* One or more of the following additional risk factors; blonde or red hair; marked freckling on the upper back; history of 3 or more blistering sunburns prior to age 20; 3 or more years of an outdoor summer job as a teenager; Actinic keratosis
* Able to give informed consent
* English speaking
* Has residential phone service
* No personal history of CMM or non-melanoma skin cancer
* No personal history of dysplastic nevi

Exclusion Criteria - FDR:

* 2 or more first degree relatives with CMM
* Has had a total cutaneous examination (TCE) in the past 3 years AND has done skin self-examination (SSE) more than once in the past year AND has a sun protection habits mean score greater than or equal to 4 (often). We are selecting a set participants who are NOT compliant with TCE and are inconsistent/minimal performers of SSE and sun protection practices.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2005-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Impact of generic print and phone counseling vs. tailored print and phone counseling interventions on the engagement in total cutaneous examination (TCE) and self-skin examination (SSE) among first degree relatives (FDRs) at increased risk for CMM. | approximately 9 months per participant

SECONDARY OUTCOMES:
Determine whether the interventions have an impact on attitudinal factors and whether these attitudinal factors mediate the expected association between the interventions and skin surveillance and sun exposure/protection. | approximately 9 months per participant

CONTACTS AND LOCATIONS:
Overall Officials: Paul Jacobsen, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Sharon L Manne, PhD, Principal Investigator — Fox Chase Cancer Center; Michael Ming, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Coups EJ, Manne SL, Jacobsen PB, Ming ME, Heckman CJ, Lessin SR. Skin surveillance intentions among family members of patients with melanoma. BMC Public Health. 2011 Nov 14;11:866. doi: 10.1186/1471-2458-11-866. PMID 22082038
- [Result] Manne S, Jacobsen PB, Ming ME, Winkel G, Dessureault S, Lessin SR. Tailored versus generic interventions for skin cancer risk reduction for family members of melanoma patients. Health Psychol. 2010 Nov;29(6):583-93. doi: 10.1037/a0021387. PMID 21090893
- [Result] Manne SL, Coups EJ, Jacobsen PB, Ming M, Heckman CJ, Lessin S. Sun protection and sunbathing practices among at-risk family members of patients with melanoma. BMC Public Health. 2011 Feb 21;11:122. doi: 10.1186/1471-2458-11-122. PMID 21338483